CLINICAL TRIAL: NCT00670735
Title: HCRN Core Data Project: Characterizing Patient Populations in the Hydrocephalus Clinical Research Network (HCRN)
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, richard holubkov, Ph.D., University of Utah
Other Study IDs: 27896; HCRN 001 (Other: HCRN Protocol Number); 1RC1NS068943-01 (NIH)
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Hydrocephalus
Keywords: Pediatric Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Hydrocephalus Clinical Research Network (HCRN) has been established by philanthropic funding to conduct multi-institutional research (clinical trials and observational studies) on pediatric hydrocephalus. In addition to philanthropic funding, the HCRN has also received an NIH NINDS Challenge Grant to support the network infrastructure which allows for the conduct of this and other network studies. The HCRN consists of multiple Clinical Centers and the Data Coordinating Center (DCC). The HCRN Core Data Project will obtain data about all neurosurgical hydrocephalus events from the network Clinical Centers, and create a database to be used by HCRN investigators. The ongoing maintenance of the Core Data Project serves two main purposes: 1) it will help investigators understand the variability, progression, and current treatment practices for hydrocephalus in children, with an ultimate goal of better guiding and assessing therapeutic intervention and providing recommendations on patient care and, 2) it will provide pilot and descriptive data necessary for hypothesis generation and study design (i.e. preliminary power analyses, recruitment projections) for studies under development by the HCRN. This multi-institutional database will be maintained throughout the lifetime of the HCRN, and may be useful for tracking trends in pediatric hydrocephalus over time. The Core Data Project will be an invaluable resource to the HCRN and will help stimulate new research protocols, identify potential need for future expansion of the network to incorporate additional patient populations, and provide a descriptive understanding of children with hydrocephalus cared for within the network.

ELIGIBILITY:
Inclusion Criteria:

Information for all neurosurgical hydrocephalus patient events will be obtained from each HCRN Clinical Center and will be placed continuously into the Core Data Project. The first calendar year will be 2008, and data collection will continue for the duration of the existence of the HCRN. Neurosurgical hydrocephalus patient events include any operation for the treatment of documented hydrocephalus including the following:

* Ventriculoperitoneal shunt
* Ventriculoatrial shunt
* Ventriculopleural shunt
* Arachnoid cyst shunts
* Subdural shunts
* Lumboperitoneal shunts
* Shunts replaced after treatment of infection
* Shunts exposed during an operations but not revised
* Endoscopic third ventriculostomies
* Ommaya reservoir(s)
* Ventricular access devices/reservoirs
* Subgaleal shunts.

Exclusion Criteria:

The following temporary cerebrospinal fluid (CSF) diversion procedures will not be included in the Core Date Project:

• External ventricular drain(s)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Hydrocephalus patients.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2008-04; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To describe the number and characteristics of neurosurgical hydrocephalus patient events to HCRN Clinical Centers such as patient demographics, etiology of hydrocephalus, diagnostic information, as well as surgical and medical management decisions. | 5+ years

SECONDARY OUTCOMES:
To provide this data to HCRN investigators to support hypothesis generation and study design development for clinical trials and observational studies to be carried out by the HCRN. | 5+ years

CONTACTS AND LOCATIONS:
Overall Officials: Jay Riva-Cambrin, MD, Study Chair — Alberta Children's Hospital; Abhaya Kulkarni, MD, PhD, Principal Investigator — Sick Children's Hospital, Toronto, Ontario; Tamara D Simon, MD, MSPH, Principal Investigator — University of Washington / Seattle Children's Hospital; Richard Holubkov, Ph.D., Principal Investigator — University of Utah
Locations (14):
- United States (11):
  - Children's Hospital of Alabama, University of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Sick Children's Hospital, Toronto, Ontario

REFERENCES:
- See also: Hydrocephalus Clinical Research Network — http://www.hcrn.org